CLINICAL TRIAL: NCT04936659
Title: Effect of Palpatory Neuromodulation of the Trigeminal Nerve for Tenderness in the Posterior Neck Musculature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Kendi Hensel, Professor, University of North Texas Health Science Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1444471
Record Dates: First submitted 2021-03-12; First posted 2021-06-23 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Neuromodulation; Neck Pain
Keywords: trigeminal nerve
MeSH Terms: conditions — Neck Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Other: neuromodulation

INTERVENTIONS:
Other: neuromodulation — Palpatory neuromodulation of the V1 and V2 branches of the trigeminal nerve where they exit onto the face.

SUMMARY:
The purpose of this study is to assess the extent to which a non-invasive, palpatory neuromodulatory protocol on the trigeminal nerve endings on the face can affect tenderness felt on the posterior neck musculature, using the Isotouch pressure sensor system.

Specific Aim 1: Subjects will see a decrease in tenderness in the posterior neck musculature.

Specific Aim 2: Subjects will show a decrease in tenderness on the trigeminal tender points found on the face.

DETAILED DESCRIPTION:
Study Instrumentation: The Isotouch sensor device and software is a passive sensor device that allows for real-time, constant visualization of pressure information. The system electronics are remote (on the packet usually worn on the wrist) and the current supports a Bluetooth data stream. The sensor has input power on the wrist and minimal microcurrent output. The pressure range for the device ranges from 0-100 pounds per square inch (PSI), although this study will only be using pressure of 0.5 to three pounds of pressure. The sensors are made of both cloth and Polyimide material. This software will be directly used in the neuromodulatory intervention as described below. The sensors will be used both for the palpatory evaluation of trigeminal tender points on the face as well as the neuromodulation portion of the protocol.

Subjects interested in the study will email the NeckPainResearch@unthsc.edu account to express their interest in participating. The co-investigators will email the subject an initial survey to answer questions about the inclusion and exclusion criteria. This survey will primarily consist of questions related to the potential participant's medical history, to best determine if they qualify for the study. If subjects qualify, they will be contacted via telephone (by the principal or a co-investigator) to schedule a time to participate in the study visit. Once a visit is scheduled, the participant will meet the investigators in a private setting either at the UNTHSC campus or other community based designated area. After the consenting process is completed, the inclusion and exclusion criteria will be re-reviewed. If the subject qualifies, they will be consented and fill out a brief questionnaire. Subjects will be verbally asked for demographic information including their age, weight, height, gender, and have their neck circumference measured by the principal investigator or a co-investigator.

After consenting, the subject will be taken to the operator (the principal or co-investigator) who will be in clinical patient room with the IsoTouch software (see diagram). The subject will lie supine on the exam table.

The operator will be wearing two IsoTouch finger sensors; one on each index finger. Non-latex coverings will be used over the IsoTouch software pressure sensors to protect the instrumentation from the natural oils of human skin, as well as the participant. The operator will palpate 1 inch posteromedial from the posterior aspect of the mastoid process (posterior neck) on each side with 3 pounds of pressure to determine if any tenderness is present, and the subject will verbally give a pain rating between 0-10. This will be referred to as the left and right cervical sites of tenderness (CSOT).

Next, using the IsoTouch finger sensor, the trigeminal nerve endings will be palpated for tenderness with 2 lbs of pressure and subjects will verbally give a pain rating on a scale of 0-10 at the following sites: V1, and V2 branches of the trigeminal nerve on the face which will be referred to as trigeminal tender points (TTPs, see below diagram). The three most tender TTPs will be documented.

Two lbs of pressure will be used on the facial sites as the anatomy is significantly different. The facial structures in general are much more superficial than the layers of musculature in the posterior neck. Therefore, the pressure will be less on the face than it is on the posterior neck musculature.

The operator will keep one monitoring sensor with minimal pressure (less than 0.5 lbs of pressure) at the CSOT while the other sensor/sensing hand applies steady pressure to each of the TTPs. The CSOT remains the same throughout the protocol and does not change sides, as it will be reevaluated when the protocol is completed.

The three most tender TTPs will be palpated with steady pressure (two lbs of pressure) for 30 seconds, as this step is the neuromodulation intervention. In the event that there are two tender points rated the same (and not zero), the investigators will repeat assessment of each trigeminal area again to be rated by the subject. If it happens that the same values are again recorded, the investigators will include both tender points in our protocol, potentially including four TTPs in the intervention. Any anomalies will be noted in the data collection. The steady pressure is continuously recorded via the pressure sensing IsoTouch pads and monitored in real time by the operator to keep it consistent with each intervention. After the TTP's have the intervention, their face will not be touched again.

After all three of the TTPs assessed to have tenderness have received the intervention, the CSOT will be rechecked with the same initial pressure (3lbs) to evaluate pain changes.

For Example, The CSOT on the right was assessed to have an 8/10 tenderness to palpation. V1R, V2R, V2L were found to have the most tenderness. In sequential order, V1R, V2R, V2L will have the neuromodulatory pulsations applied to them, and when complete, the right sided CSOT will be rechecked.

Due to the force signal drift of the ISOTOUCH, and the real-time nature of the software, the pressure/force will be monitored and adjusted accordingly to maintain the appropriate pressure/force throughout the intervention.

This neuromodulatory protocol is finished when the TTPs that were assessed to have the most tenderness each had the 30 second intervention.

The protocol will be ended immediately if any subject asks to stop, or if any significant pain or side effects develop.

ELIGIBILITY:
Inclusion Criteria:

* . Aged 18-65 2. Has posterior neck muscle discomfort 3. Has none of the following within the past 12 months:

  * traumatic brain injury
  * concussion
  * whiplash
  * dental work (cavity filling, root canal, tooth extraction, tooth implantation)
  * facial trauma
  * facial reconstruction surgery
  * diagnosis of migraine headaches with daily or weekly medication use
  * diagnosis of cluster type headaches with daily or weekly medication use 4. No neurological diagnoses, such as:

    * trigeminal neuralgia
    * facial numbness
    * paralysis of the face 5. No cervical spine issues such as:
    * Bulging disc
    * Vertebral fusion surgery
    * Vertebral disc removal surgery 6. No skin disorder of the face, neck or scalp such as:
    * Shingles/Herpes Zoster 7. Subject is able to lay supine for 15 minutes 8. Not pregnant

Exclusion Criteria:

* 1. Below the age of 18 or over the age of 65 2. Any of the following within the past 12 months:

  * traumatic brain injury
  * concussion
  * whiplash
  * dental work (cavity filling, root canal, tooth extraction, tooth implantation)
  * facial trauma
  * facial reconstruction surgery.
  * Diagnosis of migraine headaches with daily or weekly medication use
  * Diagnosis of cluster headaches with daily or weekly medication use 3. Any of the following neurologic diagnoses:

    1. trigeminal neuralgia
    2. facial numbness
    3. paralysis of the face
    4. Cervical spine issues (bulging disc, vertebral fusion, or vertebral disc removal)
    5. Skin disorders of the face, neck, or scalp such as Shingles or Herpes Zoster
    6. Pregnancy
    7. Unable to lay on back for 15 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Cervical muscle tenderness | Change from pre to immediately post intervention
  Palpatory assessment of muscle tenderness measured on a visual analog scale of 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Kendi Hensel, DO, PhD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No